CLINICAL TRIAL: NCT03083028
Title: Combined Randomised and Observational Study of Surgery for Type B Ankle Fracture Treatment
Acronym: CROSSBAT 5Y
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The University of New South Wales (Other)
Responsible Party: Principal Investigator, Rajat Mittal, Principal Investigator, The University of New South Wales
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CROSSBAT 5Y
Record Dates: First submitted 2017-03-12; First posted 2017-03-17 (Actual); Last update posted 2017-03-17 (Actual); Status verified 2017-03

CONDITIONS: Ankle Fractures
Keywords: Ankle Fracture
MeSH Terms: conditions — Ankle Fractures

STUDY DESIGN:
Intervention Model Description: Randomised Controlled Trial with an Observational Cohort
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor were masked to the treatment allocation of participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non Operative (Active Comparator): Non-Operative
  Patients who are treated non-operatively will be treated with a walking boot and allowed WBAT. Discharge from hospital will be determined by the patient walking 25m unaided by standby assistance. All patients will be reviewed between 7 and 14 days post injury with repeat x-rays by the treating surgeon.
  Interventions: Procedure: Non Operative
- Operative (Active Comparator): The specific procedure for each patient managed operatively, both in the observational study and the RCT, will be determined by the operating surgeon. Any adverse intra-operative or post-operative event will be recorded. This includes but is not limited to death, infection and neurovascular injury. Post operatively, all patients will be NWB (non weight bearing) and placed in a POP (plaster of paris) below knee cast or walking boot. Discharge from hospital will be determined by the patient walking 25m unaided by standby assistance. The treating surgeon will review the patients after 10-14 days for a wound review, removal of sutures and change of cast to a fibreglass cast or walking boot (cam walker). The patient will be WBAT (weight bearing as tolerated) for a further 4 weeks
  Interventions: Procedure: Open reduction internal fixation of the ankl

INTERVENTIONS:
Procedure: Non Operative — Patients who are treated non-operatively will be treated with a walking boot and allowed WBAT. Discharge from hospital will be determined by the patient walking 25m unaided by standby assistance. All patients will be reviewed between 7 and 14 days post injury with repeat x-rays by the treating surgeon.
  Arms: Non Operative
Procedure: Open reduction internal fixation of the ankl — The specific procedure for each patient managed operatively, both in the observational study and the RCT, will be determined by the operating surgeon. Any adverse intra-operative or post-operative event will be recorded. This includes but is not limited to death, infection and neurovascular injury. Post operatively, all patients will be NWB (non weight bearing) and placed in a POP (plaster of paris) below knee cast or walking boot. Discharge from hospital will be determined by the patient walking 25m unaided by standby assistance. The treating surgeon will review the patients after 10-14 days for a wound review, removal of sutures and change of cast to a fibreglass cast or walking boot (cam walker). The patient will be WBAT (weight bearing as tolerated) for a further 4 weeks.
  Arms: Operative

SUMMARY:
This study will determine whether operative management confers improved short and long-term outcomes for patients with isolated AO type 44-B1 distal fibula fractures when compared with non-operative management.

DETAILED DESCRIPTION:
Background:

Ankle fractures are common. Recent clinical studies have shown that there is an increasing incidence of ankle fractures. Treatments vary and there is no clear consensus of the ideal approach to type 44-B1 distal fibular fractures. They range from open reduction and internal fixation to restore anatomical alignment to wearing below-knee walking plaster for an average of six weeks.

The argument for surgical fixation is that it addresses minor displacement and possible future displacement therefore potentially preventing future arthritis. On the other hand, there are numerous complications associated with surgery.

The argument for non-operative treatment is that non-union is not a common complication. Therefore surgery can be avoided in the majority of cases avoiding the clinical risks associated with surgery.

Aim:

Primary aim: To compare, ankle function and quality of life 5 years following an isolated AO type 44-B1 distal fibula fracture minimal talar shift, between patients treated operatively and non-operatively.

Research Design: Combined Randomised and Observational Study

Methods:

Recruitment:

All consecutive patients who present to a recruiting hospital with a distal fibular fracture during the study period will be screened for eligibility. In most hospitals, all surgeons on the on-call roster will participate in the study. Consenting patients of the surgeons who have agreed to participate in the randomised arm of the trial will be invited to have their treatment randomised. Patients of surgeons involved in the observational component of the study will be invited to be included in the observational arm together with the patients who decline to be randomised, but consent to follow-up

Written, informed consent will be obtained.

Eligible patients of surgeons participating in the randomised arm will have the option of having their treatment randomised. If consent is given, the surgeon will call a central number for patient allocation that is available 24 hours per day, 7 days per week. The randomisation schedule will be prepared and administered by an external party not otherwise involved in the study. If the patient declines randomisation, treatment will be determined after surgeon-patient discussion. Eligible patients of surgeons involved in the observational arm will also have their treatment provided (operative or non-operative) as per usual surgeon practice.

Typical demographic, anthropometric and surgical details (where appropriate) will be recorded for contextual reference.

Surgical intervention:

The surgical technique for each patient managed operatively, in both the observational and randomised arms of the study, will include fixation using a plate and screws. Any adverse intra-operative or post-operative event will be recorded. This includes but is not limited to death, infection, VTE and neurovascular injury. Post-operatively, all patients will be non weight bearing and placed in a below-knee plaster cast or walking boot. Discharge from hospital will be determined by the patient's ability to walk 25 m unaided by standby assistance as determined by a physiotherapist. The treating surgeon will review the patient after 10-14 days for assessment of the wound, removal of sutures and change of cast to a fibreglass cast or walking boot (cam walker). The patient will then be allowed to WBAT (weight bearing as tolerated) for a further 4 weeks. This protocol represents usual post-operative practice for this injury, as determined through meetings with the Australian Orthopaedic Trauma Society.

Non-Operative management:

Patients who are treated non-operatively will be treated with a walking boot and allowed WBAT. Discharge from hospital will be determined as for the surgical arm. All patients will be reviewed between 7 and 14 days post injury with repeat radiographs by the treating surgeon. This represents usual non-operative treatment for this injury.

Other management decisions such as need for antibiotics, VTE prophylaxis or anaesthetic type will be as per usual care for that institution and recorded by the research team. Referral for further physiotherapy post removal of cast or boot (either study arm) will be based on the presence of overt ankle stiffness affecting gait. The use of physiotherapy (type and duration) will be noted. Specific prescription of the type of physiotherapy is not possible as patients will be free to access public and private services. Study participants will record all hospitalisations and visits to any health professional. They will be required to report the main reason for such health service occasions during the first year of follow-up period.

Outcomes will be collected and results will be reported in peer-reviewed journals after appropriate statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

- Arbeitsgemeinschaft für Osteosynthesefragen (AO) type 44-B1 fibula fracture Patients aged between 18 and 65 inclusive. No talar shift - Medial clear space less than 2mm compared with the superior clear space on anterior-posterior (AP) view of the ankle.

Closed injury No concurrent fractures/dislocations Mobilising unaided/independently pre-injury Willingness to be followed up for 12 months Able to provide informed written consent

Exclusion Criteria:

- Medically fit for general anaesthesia/surgery Dislocation on presentation Skeletally immature patients Previous trauma or surgery to the affected ankle Pregnancy Other injuries that impede mobilisation e.g. stroke, neurovascular deficit at presentation Non-English speaking

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2010-08; Primary Completion 2019-09 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
American Academy of Orthopaedic Surgeons Foot and Ankle Questionnaire | 5 years
  American Academy of Orthopaedic Surgeons Foot and Ankle Questionnaire
PCS of Short Form (SF)-12v2 | 5 years
  SF-12 version 2 Health Survey

SECONDARY OUTCOMES:
Complications | 5 years
  Late surgery Infection Neurovascular complication Mortality
MCS of Short Form (SF)-12v2 | 5 years
  SF-12 version 2 Health Survey

CONTACTS AND LOCATIONS:
Overall Officials: Rajat Mittal, BSc (Med), MBBS, MMed, MS, Principal Investigator — University of New South Wales